CLINICAL TRIAL: NCT06153914
Title: A Clinical Study of the Effectiveness of Sequential Adult Left Lateral Lobe Liver Transplantation in Patients With Hepatitis B Cirrhosis: a Single-center, Prospective, Single-arm Study
Brief Title: SALT for Patients With Hepatic Cirrhosis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LY2023-223
Record Dates: First submitted 2023-11-22; First posted 2023-12-01 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Liver Cirrhosis; Liver
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Surgical group (Experimental): This study intends to select patients with decompensated hepatitis B cirrhosis who meet the enrollment criteria and perform sequential adult left lateral lobe liver transplantation.
  Interventions: Procedure: Sequential Adult Left Lateral Liver Transplantation

INTERVENTIONS:
Procedure: Sequential Adult Left Lateral Liver Transplantation — Hemihepatectomy combined with orthotopic left lateral lobe liver transplantation is performed first, and residual liver resection is performed after the graft has grown to a sufficient functional liver volume. After the two-stage surgery, we will follow up on all subjects for one year.

SUMMARY:
Hepatitis B virus (HBV) infection is a very difficult public health problem in the world. Patients often experience the trilogy of "hepatitis-cirrhosis-liver cancer". Patients with decompensated cirrhosis may develop a variety of complications, such as portal hypertension, hypersplenism, esophageal and gastric variceal bleeding, ascites, spontaneous peritonitis, hepatic encephalopathy, etc.

Liver transplantation is the only way to cure hepatitis B cirrhosis. However, the shortage of liver donors still severely limits its development. In 2015, Line and others proposed a new surgical method, namely resection and partial liver segment 2-3 transplantation with delayed total hepatectomy (RAPID). This surgery innovatively combines auxiliary liver transplantation and ALLPS surgery, which can greatly alleviate the problem of liver donor shortage and improve the overall prognosis of the above-mentioned patients.

Our center has designed the Sequential Adult Left Lateral Liver Transplantation (SALT) procedure based on the principles of RAPID surgery and the characteristics of patients with cirrhosis. Compared with RAPID surgery, SALT surgery can dynamically monitor and regulate the blood flow of the residual liver and transplanted liver, reducing the risk caused by portal hypertension. This study will evaluate the safety and effectiveness of SALT in the treatment of post-hepatitis B cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* ①Age 18-75 years old;

  * Have a history of hepatitis B infection;

    * The imaging results are consistent with the manifestations of liver cirrhosis;

      * One of the following conditions: Meld score 15-40 points, esophageal and gastric variceal bleeding, refractory ascites, recurrent hepatic encephalopathy, hepatorenal syndrome, or hepatopulmonary syndrome; ⑤PS score 0-1 points; ⑥Sign the informed consent form.

Exclusion Criteria:

* ①Severe thrombosis or cavernous degeneration in the portal vein system, and liver transplantation is contraindicated upon evaluation;

  * Hepatic encephalopathy stage IV;

    * Pulmonary arterial hypertension (moderate to high risk, WHO grade III-IV) that does not improve after medical treatment or is assessed to have contraindications for surgery; ④Special types of anatomical variations;

      * Inability to tolerate surgical anesthesia (such as severe infection, cardiopulmonary insufficiency, cerebrovascular disease, etc.); ⑥Severe mental illness; ⑦Other reasons that the researcher believes are not suitable for participation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
survival rate | 1 month, 3 months, 6 months and 1 year post-transplant
  To explore the 1-year overall survival rate of patients with hepatitis B cirrhosis treated with SALT.

IPD SHARING:
Plan to Share IPD: No